CLINICAL TRIAL: NCT06303557
Title: Effect of ESPB on Intraoperative Remifentanil Consumption in Lumbar Spine Surgery
Brief Title: Effect of ESPB on Intraoperative Remifentanil Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2023-797
Record Dates: First submitted 2024-02-26; First posted 2024-03-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Spine Surgery; Erector Spinae Plane Block; Remifentanil Consumption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative Erector Spinae Plane Block (Active Comparator): In the preoperative period, under general anesthesia, after the linear ultrasound (US) probe will be placed 2-3 cm lateral to the L3 spinous process, 15 ml of 0.25% bupivacaine will be injected into the interfacial space below the erector spinae muscle, above the transverse process. The same ESPB procedure was performed on the other side. In total, 30 ml of 0.25% bupivacaine was administered.
  Interventions: Drug: Preoperative Erector Spinae Plane Block
- Postoperative Erector Spinae Plane Block (Active Comparator): In the postoperative period, under general anesthesia, after the linear ultrasound (US) probe will be placed 2-3 cm lateral to the L3 spinous process, 15 ml of 0.25% bupivacaine will be injected into the interfacial space below the erector spinae muscle, above the transverse process. The same ESPB procedure was performed on the other side. In total, 30 ml of 0.25% bupivacaine was administered.
  Interventions: Drug: Postoperative Erector Spinae Plane Block

INTERVENTIONS:
Drug: Preoperative Erector Spinae Plane Block — Erector spinae plane block will be performed bilaterally, under US guidance, before the surgical operation, after the induction of anesthesia, and when the patient is placed in the prone position.
  Arms: Preoperative Erector Spinae Plane Block
Drug: Postoperative Erector Spinae Plane Block — Erector spinae plane block will be performed unilaterally, under US guidance, after the surgical operation, under general anesthesia, and when the patient is placed in the prone position.
  Arms: Postoperative Erector Spinae Plane Block

SUMMARY:
In recent years, regional anesthesia techniques have also been frequently applied to patients for pain relief. Erector spinae plane block (ESPB), is among the regional anesthesia techniques frequently used in lumbar spine surgery.

General anesthesia (GA) is the main method of anesthesia for lumbar spine surgery. However, GA can only inhibit the projection system of the cortical limbic system or hypothalamic cortex. GA cannot completely block the transmission of peripheral noxious stimulus to the central nervous system and cannot effectively inhibit the intraoperative stress response. With the addition of peripheral blocks such as ESPB, lower remifentanil consumption, and more stable hemodynamics are expected by providing preemptive analgesia in patients.

As a result of all these; it was aimed to compare the intraoperative remifentanil consumption of patients who underwent preoperative ESPB in patients who will undergo lumbar spine surgery resection under GA with those who underwent postoperative ESPB.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* American Society of Anesthesiologists (ASA) physical status I-II-III
* Body mass index 18 to 30 kg/m2
* Elective lumbar disc herniation surgery

Exclusion Criteria:

* Patient refusing the procedure
* Patients who have previously undergone spinal surgery
* Chronic opioid or analgesic use
* Patients who will operate under emergency conditions
* Patients who will not undergo lumbar disc herniation surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Intraoperative remifentanil consumption | During the intraoperative period
  The amount of remifentanil that patients need to maintain anesthesia during the intraoperative period will be recorded.

SECONDARY OUTCOMES:
Mean arterial pressure | Perioperative period
  Mean arterial pressure values will be recorded before anesthesia, before surgical incision, after surgical incision at the 5th, 30th, 60th, 90th, 120th minutes, and after general anesthesia.
Heart rate | Perioperative period
  Heart rate values will be recorded before anesthesia, before surgical incision, after surgical incision at the 5th, 30th, 60th, 90th, 120th minutes, and after general anesthesia.
Pain scores | First 24 hours after surgery
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at the 1st, 2nd, 6th, 12th, and 24th hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)